CLINICAL TRIAL: NCT01391117
Title: A Phase Ib, Double-Blind, Randomized, Placebo-Controlled Trial in Genotype 1 HCV-Infected Subjects to Determine the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Repeated Doses of TMC649128 Given as Monotherapy and Given in Combination With Pegylated Interferon + Ribavirin
Brief Title: TMC649128HPC1002 - a Trial inGenotype 1 Hepatitis C Virus (HCV) - Infected Participants to Determine the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of TMC649128, Alone and Combined With Pegylated Interferon + Ribavirin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Antiviral activity was considered insufficient to warrant further clinical development of TMC649128.
Sponsor: Tibotec BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017992; TMC649128HPC1002 (Other: Tibotec-Virco Virology BVBA); NCT01532557 (obsolete NCT alias)
Record Dates: First submitted 2011-06-13; First posted 2011-07-11 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis C Virus
Keywords: TMC649128; HCV; TMC649128HPC1002; Hepatitis C; Hep C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- 010 (Experimental): TMC649128 panel 4 arm 2: 10 participants receive PegIFN a-2a/RBV in combination with TMC649128 administered q12h or q24h for 14 days. Actual dose and dose regimen (12h or 24h) is to be selected based on panels 1 2 and 3.
  Interventions: Drug: TMC649128
- 001 (Experimental): TMC649128. panel 1: 8 participants receive a q24h regimen at 1000 mg of TMC649128.
  Interventions: Drug: TMC649128.
- 002 (Placebo Comparator): placebo. panel 1: 2 participants receive placebo at a q24h regimen.
  Interventions: Drug: placebo.
- 003 (Experimental): TMC649128. panel 2 arm 1: 8 participants receive a q12h regimen of TMC649128 at a selected dose based on results of panel 1.
  Interventions: Drug: TMC649128.
- 004 (Placebo Comparator): placebo. panel 2 arm 1: 2 participants receive placebo at a q12h regimen.
  Interventions: Drug: placebo.
- 005 (Experimental): TMC649128. panel 2 arm 2: 8 participants receive a q24h regimen TMC649128 at a dose based on results of panel 1.
  Interventions: Drug: TMC649128.
- 006 (Placebo Comparator): placebo. panel 2 arm 2: 2 participants receive placebo at a q24h regimen.
  Interventions: Drug: placebo.
- 007 (Experimental): TMC649128 panel 3: 8 participants receive TMC649128. Actual dose and dose regimen (q12h or q24h) to be selected based on the results of the panels 1 and 2.
  Interventions: Drug: TMC649128
- 008 (Placebo Comparator): placebo. panel 3: 2 participants receive placebo. Actual dose and dose regimen (q12h or q24h) to be selected based on the results of the panels 1 and 2.
  Interventions: Drug: placebo.
- 009 (Placebo Comparator): placebo panel 4 arm 1: 10 participants receive PegIFN a-2a/RBV in combination with placebo administered q12h or q24h for 14 days. Actual dose and dose regimen (12h or 24h) is to be selected based on panels 1 2 and 3.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo. — panel 1: 2 participants receive placebo at a q24h regimen.
  Arms: 002
Drug: placebo. — panel 3: 2 participants receive placebo. Actual dose and dose regimen (q12h or q24h) to be selected based on the results of the panels 1 and 2.
  Arms: 008
Drug: TMC649128. — panel 2, arm 1: 8 participants receive a q12h regimen of TMC649128 at a selected dose based on results of panel 1.
  Arms: 003
Drug: placebo. — panel 2, arm 2: 2 participants receive placebo at a q24h regimen.
  Arms: 006
Drug: placebo — panel 4, arm 1: 10 participants receive PegIFN a-2a/RBV in combination with placebo, administered q12h or q24h, for 14 days. Actual dose and dose regimen (12h or 24h) is to be selected based on panels 1, 2 and 3.
  Arms: 009
Drug: TMC649128 — panel 4, arm 2: 10 participants receive PegIFN a-2a/RBV in combination with TMC649128, administered q12h or q24h, for 14 days. Actual dose and dose regimen (12h or 24h) is to be selected based on panels 1, 2 and 3.
  Arms: 010
Drug: TMC649128. — panel 2, arm 2: 8 participants receive a q24h regimen TMC649128 at a dose based on results of panel 1.
  Arms: 005
Drug: TMC649128 — panel 3: 8 participants receive TMC649128. Actual dose and dose regimen (q12h or q24h) to be selected based on the results of the panels 1 and 2.
  Arms: 007
Drug: TMC649128. — panel 1: 8 participants receive a q24h regimen at 1000 mg of TMC649128.
  Arms: 001
Drug: placebo. — panel 2, arm 1: 2 participants receive placebo at a q12h regimen.
  Arms: 004

SUMMARY:
The purpose of this study is to determine in genotype 1 Hepatitis C Virus (HCV)-infected participants, the safety, tolerability, pharmacokinetics (how the drug is absorbed in the body, how it is distributed within the body and removed from the body over time) and antiviral activity of repeated doses of TMC649128 given as monotherapy and given in combination with pegylated interferon + ribavirin. We assess the pharmacokinetic/pharmacodynamic (how the study medication affects the body) (PK/PD) relationship for antiviral activity, active metabolite and safety of TMC649128 and its metabolites. We determine the short term safety and tolerability of the co-administration of TMC649128 and pegylated interferon + ribavirin during multiple dosing for 14 days in treatment-naive genotype 1 HCV-infected participants. We explore the effect of pegylated interferon + ribavirin on the pharmacokinetics of TMC649128 during the multiple dosing for 14 days in treatment-naive genotype 1 HCV-infected participants. We also assess in a preliminary way the short term antiviral effect of the combination of TMC649128 with pegylated interferon + ribavirin during a 14-day dosing period in treatment-naive genotype 1 HCV-infected participants.

DETAILED DESCRIPTION:
TMC649128 is a nucleoside inhibitor (NI) of hepatitis C virus (HCV) polymerase in development for the treatment of chronic hepatitis C infection. Treatment-naive genotype 1 HCV-infected participants are participants who have never received (pegylated) interferon ([Peg]IFN), ribavirin (RBV) or any other approved or investigational treatment for chronic HCV infection. Treatment-experienced genotype 1 HCV-infected participants are defined as previous non-responder and relapse subjects to previous treatment regimens (IFN/RBV or PegIFN/RBV), who have never received a HCV polymerase inhibitor and HCV protease inhibitor treatment was stopped since at least one year. This study is a Phase Ib, double-blind, randomized, placebo-controlled trial in genotype 1 HCV-infected participants to determine the safety, tolerability, pharmacokinetics and antiviral activity of repeated doses of TMC649128 given as monotherapy and given in combination with pegylated interferon + ribavirin. This trial consists of 2 phases. In the first phase TMC649128 will be given as monotherapy during 10 days at different doses and dosing regimens. In the second phase TMC649128 will be administered at one selected dose regimen in combination with PegIFN a-2a/RBV for 14 days.; All dosages of TMC649128 or placebo are given orally under fed conditions.; The monotherapy phase includes 3 panels (panel 1-3) and the combination therapy phase includes 1 panel (panel 4). In panel 1, subjects are randomly assigned to receive TMC649128 at 1000 mg q24h (every 24h) (n=8) or placebo (n=2) q24h on Days 1-10. In panel 2 subjects are randomized into Arm 1 and Arm 2 and within each arm, subjects are randomly assigned to receive TMC649128 or placebo as follows: In arm 1 volunteers receive TMC649128 at a selected dose (n=8) or placebo (n=2) q12h on Days 1-10. In arm 2 volunteers receive TMC649128 at a selected dose (n=8) or placebo (n=2) q24h on Days 1-10. Panel 3: TMC649128 at a selected dose (n=8) or placebo (n=2) q12h (every 12h) OR q24h on Days 1-10 where the assignment is determined by randomization; Panel 4 volunteers are randomized into Arm 1 and Arm 2. In panel 4, arm 1, 10 volunteers receive placebo (q12h OR q24h, dosing regimen matched to Arm 2 of Panel 4) + PegIFN a-2a/RBV on Days 1-14. In Panel 4, arm 2, 10 volunteers receive TMC649128 at a selected dose (q12h OR q24h) + PegIFN a-2a/RBV on Days 1-14.; The actual dose of Panel 1 is derived from data obtained from the currently ongoing MC649128HPC1001 trial. The actual dose in Panel 2 will depend on the results of Panel 1 (total daily dose of TMC649128 administered in both arms of Panel 2 will be the same. The dose of TMC649128 of the q24h regimen in Arm 2 will be higher than the q24h dose administered in Panel 1 [1000 mg q24h]). The actual doses and dose regimens in Panels 3 and 4 will depend on the results of Panels 1 and 2 (data review meetings). Selection of doses and dose regimens in Panels 2, 3 and 4 will also depend on the data obtained from trial TMC649128HPC1001. Dosing will stay within the exposure limits. The intended doses for Panels 2 and 3 are 2000 mg or 3000 mg q12h or q24h, but may be adapted based on previous clinical data. If needed and based on the outcome of the Panel 1 results, subjects in Panel 3 may eventually receive a lower dose than in Panel 1. See detailed study description.

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic (> 6 months) genotype 1a or 1b Hepatitis C virus (HCV) infection
* Treatment-naive volunteer, meaning never received (Peg)IFN, RBV or any other approved or investigational treatment for chronic HCV infection (Panels 1, 2, 3 or 4) OR volunteer is a documented prior non-responder or relapser subject to previous treatment regimens (IFN/RBV or pegylated IFN/RBV) but has stopped this treatment at least 6 months before screening
* volunteer has never received a HCV polymerase inhibitor and HCV protease inhibitor treatment was stopped since at least one year (Panels 1, 2 or 3)
* Volunteer with HCV plasma RNA levels of > 100,000 IU/mL at screening
* Body Mass Index of 18.0 to 35.0 kg/m2
* Healthy based on a medical evaluation including medical history, physical examination, blood tests, vital signs, and electrocardiogram.

Exclusion Criteria:

* Evidence of liver cirrhosis
* Historical liver biopsy graded as liver cirrhosis or evidence for the presence of oesophageal varices or a transient elastography (Fibroscan) result of more than 14.6 kPa within 2 years prior to screening
* Evidence of decompensated liver disease defined as prior history or current evidence of ascites, hepatic encephalopathy, bleeding oesophageal or gastric varices
* Evidence of renal dysfunction, documented by an estimated creatinine clearance below 70 mL/min
* Evidence of any other cause of significant liver disease in addition to hepatitis C, this may include but is not limited to hepatitis B, drug- or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, non-alcoholic steatohepatitis, or primary biliary cirrhosis
* Volunteer with diagnosed or suspected hepatocellular carcinoma
* Volunteer receiving or having received any treatment for HCV during the 6 months before screening
* Volunteer coinfected with Human Immunodeficiency Virus-1 (HIV-1) or HIV-2, or hepatitis A or B virus infection, or clinically active tuberculosis at study screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in the steady-state plasma concentrations of TMC649128. | From baseline up to Day 80 per panel (panel 1 + panel 2 + panel 3).
Change in the steady-state plasma concentrations of TMC649128 following co-administration with pegylated interferon + ribavirin. | From baseline up to day 84 (panel 4).
Viral load decreases and/or changes of viral load from baseline (HCV RNA copies/ml) (PK/PD). | For monotherapy from baseline up to Day 80 per panel (panel 1 + panel 2 + panel 3) and for combination therapy from baseline up to day 84 (panel 4).
Number of participants with adverse events as a measure of safety and tolerability - TMC649128 as monotherapy and when co-administered with pegylated interferon + ribavirin. | For monotherapy from baseline up to Day 80 per panel (panel 1 + panel 2 + panel 3) and for combination therapy from baseline up to day 84 (panel 4).

SECONDARY OUTCOMES:
Antiviral activity (HCV RNA levels) of TMC649128 as monotherapy and when co-administered with pegylated interferon + ribavirin. | For monotherapy from baseline up to Day 80 per panel (panel 1 + panel 2 + panel 3) and for combination therapy from baseline up to day 84 (panel 4)
Antiviral activity (viral breakthrough) of TMC649128 as monotherapy and when co-administered with pegylated interferon + ribavirin. | For monotherapy from baseline up to Day 80 per panel (panel 1 + panel 2 + panel 3) and for combination therapy from baseline up to day 84 (panel 4).

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA
Locations (3):
- Zuidlaren, Netherlands
- Poland (2):
  - Krakow
  - Warsaw